CLINICAL TRIAL: NCT06892730
Title: Safety and Efficacy of TEVAR Combined With Long Bare-metal Stents in the Intervention of ATBAD: a Prospective and Cohort Study
Brief Title: Safety and Efficacy of TEVAR Combined With Long Bare-metal Stents in the Intervention of ATBAD
Acronym: SAFE-COVER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yan'an Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YAYY-2025-001; 82460098 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-03-15; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Aortic Dissection Type B
Keywords: ATBAD; TEVAR; Extension; Long bare metal scaffolding devices

STUDY DESIGN:
Intervention Model Description: Single Group Assignment: All enrolled subjects receive uniform intervention protocol (TEVAR combined with long bare-metal stent intervention)
Masking Description: Open-label design: Participants, operators and assessors are unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carstor® 70-240mm, AnkuraTMⅡ60-200mm, WeFlow-TbranchTM and Fabulous® Device Surgical Implant (Experimental): Subjects with acute type B aortic dissection were treated with an endovascular procedure using the Carstor® 70-240mm, AnkuraTMⅡ60-200mm, WeFlow-TbranchTM 160-240mm Thoracic Aortic Endoprosthesis and the Fabulous® 45-150mm long big bare stent via femoral artery access. (Permanent implant)
  Interventions: Device: Hybrid TEVAR combined with long bare-metal stent intervention

INTERVENTIONS:
Device: Hybrid TEVAR combined with long bare-metal stent intervention — - Primary TEVAR: Primary TEVAR: Employ Carstor® 70-240mm, AnkuraTMⅡ60-200mm, WeFlow-TbranchTM 160-240mm endograft deployed with ≥2cm proximal landing zone coverage.
  Concurrent bare-stenting: Post-TEVAR femoral access deployment of Fabulous® (45-150mm) long bare-metal stent with:
  Proximal overlap ≥3cm with TEVAR graft. Distal extension 2-6cm below renal artery plane. Maximum distal limit: above iliac bifurcation.
  - Intraprocedural angiography with spinal reference mapping guides precise stent positioning relative to visceral arteries and infrarenal aorta.

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of the TEVAR combined with extended bare-metal stenting (distal landing zone ≥2 cm below renal arteries) in patients with acute complicated type B aortic dissection (ATBAD).

Additionally, to prevent postoperative true lumen hypoperfusion in residual thoracoabdominal aortic dissection (visceral zone, infrarenal aorta, and iliac arteries) and persistent ischemic manifestations in visceral and lower extremity arteries post-endovascular repair, extended bare-metal stents are deployed to maintain adequate distal true lumen patency. This strategy ensures perfusion to visceral branches and lower limbs while preparing for future complete endovascular aortic repair.

DETAILED DESCRIPTION:
Stanford type B aortic dissection (TBAD) accounts for 25-40% of all aortic dissections, characterized by acute onset, rapid progression, and high mortality, representing a critical cardiovascular emergency. While thoracic endovascular aortic repair (TEVAR) remains the standard intervention for TBAD, its benefits on true lumen remodeling and false lumen thrombosis are primarily limited to the stent-graft covered segment. Distal to the stent-graft, persistent re-entry tears in thoracoabdominal arteries convert preoperative exit sites into new entry points. Although TEVAR improves true lumen perfusion distal to the stent-graft, remodeling efficacy remains suboptimal, particularly in cases with preoperative true lumen collapse where post-TEVAR true lumen dimensions remain critically compressed by large false lumen volumes. Currently deployed stent-grafts typically measure 15-20 cm in length. Conventional TEVAR requires ≥1.5 cm proximal healthy aortic segment as landing zone to prevent retrograde type A dissection (RTAD) and ensure stability. For patients with inadequate proximal landing zones (<1.5 cm), advanced techniques including branched stent-grafts, fenestrations, and parallel grafting have enabled TEVAR implementation even with ≤0.5 cm landing zones, facilitated by evolving device technologies and operator expertise. The "TEVAR+bare-stent" hybrid approach theoretically enhances aortic remodeling through reduced radial force. However, standard TEVAR typically deploys single stent-grafts at the proximal descending aortic tear. Extended stent-graft coverage beyond celiac axis level risks visceral artery occlusion, making maintenance of distal organ and limb perfusion an enduring challenge. Moreover, residual distal thoracoabdominal dissection carries risks of false lumen aneurysmal degeneration and rupture, particularly >5 years post-TEVAR. Secondary interventions for chronic residual dissections are complicated by intimal calcification from prolonged false lumen hypertension, combined with chronic hypoxia and inflammation that compromise aortic wall integrity. Persistent false lumen expansion and rupture in residual thoracoabdominal dissection are observed in 23-35% of conventional TEVAR cases, particularly affecting young-to-middle-aged patients with suboptimal blood pressure control beyond 5-year follow-up. Technical challenges in secondary visceral branch reconstruction further compromise long-term quality of life. Therefore, post-endovascular true lumen remodeling in thoracoabdominal segments warrants particular attention, as aortic remodeling constitutes a crucial determinant of therapeutic success beyond procedural technique alone.

This study aims to validate the feasibility and safety of proximal stent-graft plus extended distal bare-metal stenting in thoracoabdominal aorta, compare its efficacy with conventional TEVAR, and characterize its impacts on aortic remodeling and subsequent visceral/distal arterial reconstruction. We anticipate this research will provide critical clinical evidence for managing residual thoracoabdominal dissection after acute TBAD repair.

Using imaging-based analysis and clinical follow-up, this study will compare: (1) conventional TEVAR vs. (2) hybrid proximal stent-graft + extended distal bare-stent strategies in terms of morphological remodeling, adverse events, and long-term outcomes. The findings may elucidate differential impacts on aortic reconstruction and visceral/iliac revascularization, offering evidence-based guidance for managing distal dissection in acute TBAD.

ELIGIBILITY:
Inclusion Criteria:

* ≧18 years old, ≦80 years old;
* Acute phase with a course of disease ≦14 days;
* CTA confirmed diagnosis of active dissection type B in accordance with the Stanford classification in the ESC guidelines, and requiring TEVAR surgery;
* For patients with acute non-type A and non-type B aortic dissection involving the left subclavian artery: current technologies (such as fenestration, single branch, chimney, etc.) can be used to solve the reconstruction of the left subclavian artery;
* The distal end of the dissection exceeds the renal artery plane;
* Signed informed consent (emergency waiver applicable), with primary intervention using CTAG devices. Adjunctive procedures may include LSA revascularization, percutaneous fenestration, aortic/peripheral stenting, surgical fenestration, or bypass grafting.
* Medical record completeness >90% with mandatory CTA data;
* Protocol compliance including follow-up adherence

Exclusion Criteria:

* Dissection termination above renal arteries;
* Major aortic surgery within 30 days prior (except LSA revascularization);
* Iliofemoral stenosis/angulation precluding endovascular access;
* Non-diagnostic CTA image quality;
* Indeterminate symptom onset time;
* Traumatic TBAD, intramural hematoma, or penetrating aortic ulcer;
* Complete thoracic aortic thrombosis pre-TEVAR;
* Re-intervention within 12 months post-TEVAR for non-aortic indications;
* Renal failure: Baseline serum creatinine >2.5 mg/dL (high-risk for contrast nephropathy);
* Known device material hypersensitivity;
* Systemic infection increasing endograft infection risk;
* Evidence of aortic infection;
* Connective tissue disorders (e.g., Marfan syndrome);
* Bowel necrosis from visceral ischemia;
* Participation in other device/drug trials within 1 year;
* Moribund status: ASA class 5 with <24h life expectancy;
* Refractory shock (SBP <90 mmHg);
* Pregnancy or lactation;
* Active substance abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality | 30 days post-intervention
  30-day all-cause mortality
Ratio of increase in aortic true lumen (%) | 1 month, 6 months, 12 months after surgery
  Ratio of increase in aortic true lumen(%) including three parameters:
  1. Diameter measurement (unit: mm): The total aortic diameter was obtained based on the 2020 SVS/STS reporting standards, and then the specific values of the true lumen diameter and false lumen diameter were obtained as a percentage of the straight line between the two lumens.
  2. Area measurement (unit: mm2): The aortic false lumen area = the true and false lumen area - the true lumen area on the same measurement plane.
  3. The change ratio (%) of true lumen diameter (mm) and area (mm2):
  Definition:
  Postoperative true lumen diameter increase ratio: (postoperative - preoperative) / preoperative*100% True lumen diameter increase ratio after follow-up: (current follow-up - last follow-up) / last follow-up*100% Postoperative true lumen area increase ratio: (postoperative - preoperative) / preoperative*100% True lumen area increase ratio after follow-up: (current follow-up - last follow-up) / last follow-up area*100%

SECONDARY OUTCOMES:
Aortic rupture incidence | 1 month, 6 months, 12 months after surgery
  Aortic rupture incidence
Device-related complications | 1 month, 6 months, 12 months after surgery
  * endoleak, spinal ischemia, organ failure
  * Classification and incidence rates
False lumen thrombosis grading | 1 month, 6 months, 12 months after surgery
  1. Complete: No contrast enhancement
  2. Partial: Partial contrast flow with thrombus
  3. Patent: Full contrast opacification

CONTACTS AND LOCATIONS:
Overall Officials: Xunqiang Prof. Liu, M.D., Principal Investigator — Yan'an Affiliated Hospital of Kunming Medical University
Locations (1):
- Yan'an Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rong D, Ge Y, Liu J, Liu X, Guo W. Combined proximal descending aortic endografting plus distal bare metal stenting (PETTICOAT technique) versus conventional proximal descending aortic stent graft repair for complicated type B aortic dissections. Cochrane Database Syst Rev. 2019 Oct 30;2019(10):CD013149. doi: 10.1002/14651858.CD013149.pub2. PMID 31684692
- [Background] Fattori R, Montgomery D, Lovato L, Kische S, Di Eusanio M, Ince H, Eagle KA, Isselbacher EM, Nienaber CA. Survival after endovascular therapy in patients with type B aortic dissection: a report from the International Registry of Acute Aortic Dissection (IRAD). JACC Cardiovasc Interv. 2013 Aug;6(8):876-82. doi: 10.1016/j.jcin.2013.05.003. PMID 23968705
- [Background] Nienaber CA, Kische S, Zeller T, Rehders TC, Schneider H, Lorenzen B, Bunger C, Ince H. Provisional extension to induce complete attachment after stent-graft placement in type B aortic dissection: the PETTICOAT concept. J Endovasc Ther. 2006 Dec;13(6):738-46. doi: 10.1583/06-1923.1. PMID 17154712